CLINICAL TRIAL: NCT01804842
Title: A Randomized, Crossover Study Assessing the Effect of EFB0027 on Plasma Glucose and Pharmacokinetics in Subjects With Type 2 Diabetes Mellitus
Brief Title: Assessing the Effect of Met DR on Plasma Glucose and PK in Subjects With T2DM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LCRM104
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 500 mg Met DR BID (Active Comparator): Two doses of 500 mg metformin delayed-release
  Interventions: Drug: Met DR
- 1000 mg Met DR qAM (Experimental): One dose of 1000 mg metformin delayed-release in the morning
  Interventions: Drug: Met DR
- 1000 mg Met DR qPM (Experimental): One dose of 1000 mg metformin delayed-release in the evening
  Interventions: Drug: Met DR

INTERVENTIONS:
Drug: Met DR — metformin delayed-release tablets
  Other Names: EFB0027

SUMMARY:
This study compared the effects of delayed-release metformin (Met DR, EFB0027) administered once daily in the morning (qAM), administered once daily in the evening (qPM), and administered twice daily (BID) on circulating glucose concentrations and metformin pharmacokinetics (PK) in subjects with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 (inclusive) years old at Visit 1 (Screening)
2. Was diagnosed with type 2 diabetes mellitus with

   * HbA1c between 6.0 to 9.5% (inclusive) for subjects managing their diabetes with:

     i. Diet and exercise alone, or ii. A stable regimen (minimum of 2 months at Visit 1) of metformin alone, or iii. A stable regimen (minimum of 2 months at Visit 1) of DPP-4 inhibitor alone OR
   * HbA1c between 6.0 to 8.5% (inclusive) for subjects managing their diabetes with a stable (minimum of 2 months at Visit 1) combination regimen of metformin and DPP-4 inhibitors
3. Had normal renal function with an estimated glomerular filtration rate (eGFR) ≥90 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease (MDRD) equation
4. Body mass index (BMI) of 25.0 to 40.0 kg/m^2 (inclusive) at Screening
5. Male, or if female and met all of the following criteria:

   * Not breastfeeding
   * Negative pregnancy test result (human chorionic gonadotropin, beta subunit) at Visit 1 (Screening) (not applicable to hysterectomized females)
   * Surgically sterile, postmenopausal, or if of childbearing potential, practiced and was willing to continue to practice appropriate birth control during the entire duration of the study
6. Had a physical examination with no clinically significant abnormalities as judged by the investigator
7. Ability to understand and willingness to adhere to protocol requirements
8. If on chronic thyroid pharmacologic therapy, the dose must have been stable for at least 3 months prior to Visit 1 (Screening), and must have thyroid-stimulating hormone (TSH) test result in normal range at Visit 1 (Screening)

Exclusion Criteria:

1. Had a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

   * Hepatic disease
   * Renal disease
   * Gastrointestinal disease
   * Endocrine disorder except diabetes
   * Cardiovascular disease
   * Central nervous system diseases
   * Psychiatric or neurological disorders
   * Organ transplantation
   * Chronic or acute infection
   * Orthostatic hypotension, fainting spells or blackouts
   * Allergy or hypersensitivity
2. Had any chronic disease requiring medication that was adjusted in the past 90 days (subjects could take acute intermittent over-the-counter medications such as Tylenol, if needed)
3. Had any drug treatment that affects gastric pH (prescription or over-the-counter), including any antacids or medications such as Rolaids or Pepcid within 2 days of Visit 1 (Screening)
4. Had major surgery of any kind within 6 months of Visit 1 (Screening)
5. Had received a blood transfusion within 6 months of Visit 1 (Screening)
6. Had a history of >5 kg weight change within 3 months of Visit 1 (Screening)
7. Had clinical laboratory test (clinical chemistry, hematology, or urinalysis) abnormalities other than those expected in subjects with type 2 diabetes and judged by the investigator to be clinically significant at Visit 1 (Screening)
8. Had a physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study
9. Abused drugs or alcohol or had a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures
10. Had donated blood within 3 months of the date of the first dose of randomized study medication, or was planning to donate blood during the study
11. Used insulin within 3 months of Visit 1 (Screening)
12. Had received GLP-1 receptor agonists and/or thiazolidinedione treatment within 6 months of Visit 1 (Screening)
13. Had known intolerance to metformin
14. Had received any investigational drug within 2 months (or five half-lives of the investigational drug, whichever was greater) of Visit 1 (Screening)
15. Had known allergies or hypersensitivity to any component of study treatment
16. Was employed by Elcelyx Therapeutics, Inc. (that is an employee, temporary contract worker, or designee of the company)
17. Smoked more than 10 cigarettes per day, 3 cigars per day, 3 pipes per day, used more than 1 can of smokeless tobacco per week, or used a combination of tobacco products that approximate nicotine doses equivalent to 10 cigarettes per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion

REFERENCES:
- [Background] Buse JB, DeFronzo RA, Rosenstock J, Kim T, Burns C, Skare S, Baron A, Fineman M. The Primary Glucose-Lowering Effect of Metformin Resides in the Gut, Not the Circulation: Results From Short-term Pharmacokinetic and 12-Week Dose-Ranging Studies. Diabetes Care. 2016 Feb;39(2):198-205. doi: 10.2337/dc15-0488. Epub 2015 Aug 18. PMID 26285584
- [Background] DeFronzo RA, Buse JB, Kim T, Burns C, Skare S, Baron A, Fineman M. Once-daily delayed-release metformin lowers plasma glucose and enhances fasting and postprandial GLP-1 and PYY: results from two randomised trials. Diabetologia. 2016 Aug;59(8):1645-54. doi: 10.1007/s00125-016-3992-6. Epub 2016 May 23. PMID 27216492

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: ABC; Sequence 2: BCA; Sequence 3: CAB: Treatment A = 1000 mg Met DR qAM Treatment B = 1000 mg Met DR qPM Treatment C = 500 mg Met DR BID
Period: Overall Study
Arm/Group | Sequence 1: ABC | Sequence 2: BCA | Sequence 3: CAB
Started | 9 | 8 | 9
Completed Treatment A | 9 | 6 | 8
Completed Treatment B | 8 | 8 | 8
Completed Treatment C | 7 | 7 | 9
Completed | 6 | 6 | 8
Not Completed | 3 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-Compliance | 1 | 1 | 0
Not completed — Personal Reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: ABC | Sequence 2: BCA | Sequence 3: CAB | Total
Number analyzed (Participants) | 9 | 8 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.73) | 51.9 (13.47) | 49.7 (8.49) | 50.9 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 16
  Male | 3 | 2 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 5 | 18
  Not Hispanic or Latino | 2 | 2 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (3.73) | 31.6 (3.93) | 30.7 (1.58) | 31.5 (3.17)
Diabetes Management [Number; unit: participants]
  Diet and Exercise Only | 1 | 4 | 2 | 7
  Metformin Alone | 7 | 3 | 7 | 17
  Metformin and DPP-4 Inhibitors | 1 | 1 | 0 | 2
Fasting Serum Glucose [Mean (Standard Deviation); unit: mg/dL] | 161.2 (29.94) | 177.6 (84.17) | 165.0 (54.02) | 167.6 (57.04)
HbA1c [Mean (Standard Deviation); unit: %] | 7.34 (1.038) | 7.13 (1.107) | 7.36 (1.022) | 7.28 (1.017)

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-24) of Plasma Metformin
Description: AUC (0-24) = Area under the curve from the start time of the standardized dinner (0 h) to 24 hours after the standardized dinner. Study medication was administered at t = 0 hours for Treatments B and C and at t = 12 hours for Treatments A and C.
Time Frame: Times points to create the AUC (0-24) were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours relative to the start time of the standardized dinner.
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: ng*h/mL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR qAM | 1000 mg Met DR qPM
Number analyzed (Participants) | 12 | 12 | 12
ng*h/mL | 7771 (619) | 5559 (433) | 7757 (604)
Statistical Analysis 1: Comparison: 1000 mg Met DR qAM vs 1000 mg Met DR qPM; 1000 mg Met DR qPM is the denominator for the % ratio of least squares (LS) means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0018, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 71.7, 90% CI 2-sided [61.14 to 84.01]
Statistical Analysis 2: Comparison: 500 mg Met DR BID vs 1000 mg Met DR qAM; 500 mg Met DR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0020, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 71.5, 90% CI 2-sided [60.85 to 84.09]
Statistical Analysis 3: Comparison: 500 mg Met DR BID vs 1000 mg Met DR qPM; 500 mg Met DR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.9844, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 99.8, 90% CI 2-sided [84.91 to 117.33]

2. Primary Outcome: Cmax of Plasma Metformin
Description: Cmax = maximum response from the start time of the standardized dinner (0 h) to 24 hours after the standardized dinner. Study medication was administered at t = 0 hours for Treatments B and C and at t = 12 hours for Treatments A and C.
Time Frame: Times points to determine Cmax were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours relative to the start time of the standardized dinner.
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR qAM | 1000 mg Met DR qPM
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 780 (71.7) | 868 (79.8) | 1035 (95.2)
Statistical Analysis 1: Comparison: 1000 mg Met DR qAM vs 1000 mg Met DR qPM; 1000 mg Met DR qPM is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.1595, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 83.8, 90% CI 2-sided [68.10 to 103.23]
Statistical Analysis 2: Comparison: 500 mg Met DR BID vs 1000 mg Met DR qAM; 500 mg Met DR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.3867, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 111.3, 90% CI 2-sided [90.37 to 136.99]
Statistical Analysis 3: Comparison: 500 mg Met DR BID vs 1000 mg Met DR qPM; 500 mg Met DR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0294, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 132.7, 90% CI 2-sided [107.78 to 163.39]

3. Primary Outcome: AUC (0-24) of Plasma Glucose
Description: as for outcome 1
Time Frame: Times points to create the AUC (0-24) were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.75, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 18.5, 19, 19.5, 20, 21, 22, 23, and 24 hours relative to the time of the standardized dinner.
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: mg*h/dL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR qAM | 1000 mg Met DR qPM
Number analyzed (Participants) | 12 | 12 | 12
mg*h/dL
  Pre-Treatment | 4668 (581) | 4947 (615) | 4961 (617)
  On-Treatment | 4438 (552) | 4503 (560) | 4509 (561)
Statistical Analysis 1: Comparison: 1000 mg Met DR qAM; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0028, ANOVA; Treatment, sequence, period, status (on-/pre-treatment) and treatment*status as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 91.0, 95% CI 2-sided [85.70 to 96.67]
Statistical Analysis 2: Comparison: 1000 mg Met DR qPM; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0024, ANOVA; [statistical method as in outcome 3, analysis 1]; % Ratio of LS Means = 90.9, 95% CI 2-sided [85.58 to 96.53]
Statistical Analysis 3: Comparison: 500 mg Met DR BID; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0992, ANOVA; [statistical method as in outcome 3, analysis 1]; % Ratio of LS Means = 95.1, 95% CI 2-sided [89.54 to 100.99]

4. Primary Outcome: Rmax (0-24) of Plasma Glucose
Description: Rmax (0-24) = maximum response from the start time of the standardized dinner (0 h) to 24 hours after the standardized dinner. Study medication was administered at t = 0 hours for Treatments B and C and at t = 12 hours for Treatments A and C.
Time Frame: Times points to determine Rmax were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.75, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 18.5, 19, 19.5, 20, 21, 22, 23, and 24 hours relative to the start time of the standardized dinner.
Population: Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR qAM | 1000 mg Met DR qPM
Number analyzed (Participants) | 12 | 12 | 12
mg/dL
  Pre-Treatment | 279 (29.9) | 290 (31.1) | 302 (32.4)
  On-Treatment | 263 (28.2) | 262 (28.1) | 273 (29.4)
Statistical Analysis 1: Comparison: 1000 mg Met DR qAM; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0006, ANOVA; [statistical method as in outcome 3, analysis 1]; % Ratio of LS Means = 90.4, 95% CI 2-sided [85.55 to 95.56]
Statistical Analysis 2: Comparison: 1000 mg Met DR qPM; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0007, ANOVA; [statistical method as in outcome 3, analysis 1]; % Ratio of LS Means = 90.5, 95% CI 2-sided [85.65 to 95.67]
Statistical Analysis 3: Comparison: 500 mg Met DR BID; Pretreatment value is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0389, ANOVA; [statistical method as in outcome 3, analysis 1]; % Ratio of LS Means = 94.3, 95% CI 2-sided [89.24 to 99.69]

ADVERSE EVENTS:
Time Frame: Approximately 36 to 91 days depending on the number of days between the start of Visit 1 and Visit 2 and the number of washout days between the treatment periods.
Arm/Group | 1000 mg Met DR qAM | 1000 mg Met DR qPM | 500 mg Met DR BID
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 6/23 | 5/24 | 7/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg Met DR qAM (N=23) | 1000 mg Met DR qPM (N=24) | 500 mg Met DR BID (N=23)
Palpitations (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Breath Odour (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 1
Thirst (General disorders) | 0 | 1 | 0
Vessel Puncture Site Bruise (General disorders) | 0 | 1 | 0
Vessel Puncture Site Pain (General disorders) | 1 | 0 | 2
Vessel Puncture Site Swelling (General disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urine Odour Abnormal (Renal and urinary disorders) | 1 | 0 | 1
Pruritus Genital (Reproductive system and breast disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.